

June 21, 2023

# To: ClinicalTrials.gov

This is a cover page to the redacted clinical protocol for APN-006 Phase 2, Randomized, 3-Period, Placebo-Controlled Crossover Study to Evaluate the Efficacy and Safety in Obstructive Sleep Apnea of AD036 versus Placebo or Atomoxetine.

The APN-006 clinical protocol is associated with NCT 04445688.

The following proprietary information was redacted from the clinical protocol for APN-006:

• IND number

#### Sincerely,

DocuSigned by:

Janu Brillain

Signer Name: Jeanne Brittain
Signing Reason: I am the author of this document
Signing Time: 6/21/2023 | 11:04:09 AM EDT

64569C0C62E54A318E0B2CE236F2917C

Jeanne Brittain Director, Program Management

# **Title Page**

**Protocol Title:** Phase 2, Randomized, 3-Period, Placebo-Controlled Crossover Study to Evaluate the Efficacy and Safety in Obstructive Sleep Apnea of AD036 versus Placebo or Atomoxetine

**Protocol Number:** APN-006

**Compound Number:** AD036

**Short Title:** AD036 Crossover Study

**Sponsor Name and Legal Registered Address:** 

Apnimed, Inc.

20 Holyoke Street

Cambridge, MA 02138

Regulatory Agency Identifying Number: IND

**Approval Date:** 15 September 2020

Version: 3.0

Date and Version of Previous Protocol: 13 April 2020, Version 2.0

# **Sponsor Signatory:**

Ronald Farkas, MD, PhD

Chief Medical Officer

15 Sept 2020

# **Table of Contents**

| 1 | Protocol Summary | 5 |
|-----|---------------------------------------|----|
| 1.1 | Synopsis | 5 |
| 1.2 | Schedule of Activities (SoA) | 6 |
| 2 | Introduction | 7 |
| 2.1 | | |
| 2.2 | Background | 7 |
| 2.2 | 7.1 Obstructive Sleep Apnea | 7 |
| 2.2 | 2.2 Unmet Medical Need | 8 |
| 2.2 | 2.3 Biological Rationale | 8 |
| 3 | Endpoints | 9 |
| 4 | Study Design | 9 |
| 4.1 | Overall Design | 9 |
| 4.2 | Scientific Rationale for Study Design | 11 |
| 4.3 | Justification for Dose | 11 |
| 4.4 | End of Study Definition | 11 |
| 5 | Study Population | 12 |
| 5.1 | | |
| 5.2 | Exclusion Criteria | 13 |
| 5.3 | Meals and Dietary Restrictions | 15 |
| 5.4 | • | |
| 5.5 | • | |
| 6 | Study Treatment | 15 |
| 6.1 | · | |
| 6.2 | • | |
| 6.3 | | |
| 6.4 | | |
| 6.5 | J I | |
| 6.6 | | |
| 7 | Discontinuation of Study Treatment | |
| 7.1 | | |
| 7.1 | 11 0 | |
| 7.2 | 1 11 0 | |
| 7.3 | • | |
| 8 | Study Assessments and Procedures | |
| 8.1 | • | |

| 8.2 | Safety Assessments | 21 |
|---|---|---|
| 8.3 | Adverse Events and Serious Adverse Events | 21 |
| 8.3.1 | Time Period and Frequency for Collecting AE and SAE Information | 21 |
| 8.3.2 | Method of Detecting AEs and SAEs | 22 |
| 8.3.3 | Follow-up of AEs and SAEs | 22 |
| 8.3.4 | Regulatory Reporting Requirements for SAEs | 22 |
| 8.3.5 | Pregnancy | 23 |
| 8.4 | Treatment of Overdose | 23 |
| 8.5 | Pharmacokinetics | 23 |
| 9 St | tatistical Considerations and Sample Size Determination | 24 |
| 9.1 | Populations for Analyses | 24 |
| 10 Sı | upporting Documentation and Operational Considerations | 25 |
| 10.1 | Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | 25 |
| 10.1.1 | Regulatory and Ethical Considerations | 25 |
| 10.1.2 | P. Financial Disclosure | 26 |
| 10.1.3 | Informed Consent Process | 26 |
| 10.1.4 | Data Protection | 27 |
| 10.1.5 | Dissemination of Clinical Study Data | 27 |
| 10.1.6 | 5 Data Quality Assurance | 27 |
| 10.1.7 | Source Documents | 28 |
| 10.1.8 | Study and Site Closure | 29 |
| 10.1.9 | Publication Policy | 29 |
| 10.1.1 | 10 Protocol Approval and Amendment | 29 |
| 10.1.1 | Il Liability and Insurance | 30 |
| 10.2 | Appendix 2: Clinical Laboratory Tests | 30 |
| Table | 2: Protocol-Required Safety Laboratory Assessments | 31 |
| 10.3 | Appendix 3: AE Definitions and Procedures for Recording, Evaluating, Follow-up, a | |
| | Reporting | |
| 10.4 | Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information | |
| 10.5 | Appendix 5: List of Abbreviations | 42 |
| 11 R | eferences | 44 |

# 1 Protocol Summary

# 1.1 Synopsis

**Protocol Title:** Phase 2, Randomized, 3-Period, Placebo-Controlled Crossover Study to Evaluate the Efficacy and Safety in Obstructive Sleep Apnea of AD036 versus Placebo or Atomoxetine

**Sponsor Study No.:** APN-006

Phase: 2

Sponsor: Apnimed, Inc.

#### **Rationale:**

AD036 is a new fixed-dose combination of atomoxetine and oxybutynin being developed for the treatment of obstructive sleep apnea (OSA). Study APN-006 is designed to confirm and extend safety and efficacy findings from the Study APN-002, a Phase 2 study of AD036 in OSA.

#### **Overall Design:**

Patients who participated in Study APN-002 are eligible for enrollment, as are new patients who meet enrollment criteria. A total of 54 Patients with baseline characteristics that predict increased responsiveness to AD036 (based on Study APN-002 findings), will be planned for enrollment.

The study is a three-period single-dose randomized crossover design in which patients will undergo overnight home sleep apnea testing (HSAT) with dosing of one of the following 3 treatments:

- Atomoxetine 80 mg + oxybutynin 5 mg
- Atomoxetine 80 mg + placebo
- Placebo + placebo

A 1-week minimum washout period will occur between each of the 3 crossover HSAT nights. The primary hypothesis is that the AD036 combination of atomoxetine and oxybutynin is superior to placebo on apnea hypopnea index (AHI). Superiority of the AD036 combination to atomoxetine is a key secondary efficacy endpoint.

#### **Number of Participants:**

A total of 54 participants are planned for enrollment.

#### **Study Duration:**

The overall study duration will be up to 10 weeks, as follows:

- Screening, up to 4 weeks;
- 3-period crossover, approximately 5 weeks;
- End of study evaluation, 1 week after end of crossover period

# **Schedule of Activities (SoA)**

Table 1 **Schedule of Activities** 

| | | 3-Period Crossover at Home | | | | Iome | | T. 1. 46. 1 | |
|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screen-<br>ing | HSAT<br>1 | Wash-<br>out <sup>2</sup> | HSAT<br>2 | Wash-<br>out | HSAT<br>3 | Wash-<br>out | End of Study<br>Evaluation <sup>1</sup> | Notes |
| Trial Day/Duration | Up to 4 weeks | Up to 5 weeks | | | | 1 week post crossover period | | | |
| Informed consent | X | | | | | | | | |
| Enrollment criteria | X | | | | | | | | |
| History and Physical | X | | | | | | | | Includes vital signs and weight |
| 12-lead ECG | X | | | | | | | | |
| Clinical laboratory and<br>serum pregnancy test<br>(WOCBP only) | X | | | | | | | | CYP2D6 test only at Screening and only for patients not previously screened in Study APN-002 |
| Drugs of abuse | X | | | | | | | | |
| Instruct and remotely oversee HSAT use | X <sup>3</sup> | X | | X | | X | | | |
| Randomization | | X | | | | | | | Occurs after enrollment criteria met, prior to HSAT 1 |
| Dispense study drug | | X | | X | | X | | | |
| HSAT | $X^3$ | X <sup>4</sup> | | X | | X | | | HSAT device provided prior to each HSAT night |
| Study drug dosing | | X | | X | | X | | | Dose at lights out; site verifies dosing remotely |
| AE/SAE monitoring | X | X | X | X | X | X | X | X | |
| Prior/concomitant medication monitoring | X | X | X | X | X | X | X | X | |

Abbreviations: AE = adverse event; HSAT = home sleep apnea test; QHS = taken at bedtime; SAE = serious adverse event; WOCBP = women of childbearing potential.

<sup>&</sup>lt;sup>1</sup> Can be conducted remotely

<sup>&</sup>lt;sup>2</sup> Each washout period is at least 7 days
<sup>3</sup> Screening HSAT only for patients without prior qualifying sleep study, and only after other study enrollment criteria confirmed as met. Screening HSAT is conducted by site and reviewed by central reading center but the investigator is responsible for confirming patient eligibility.

<sup>&</sup>lt;sup>4</sup> Remote instruction on use of HSAT and drug dosing confirmation provided by study site for each HSAT night

# 2 Introduction

# 2.1 Study Rationale

AD036 is a new fixed-dose combination of atomoxetine and oxybutynin being developed for the treatment of obstructive sleep apnea (OSA). Study APN-006 is designed to confirm and extend safety and efficacy findings from the Phase 2 Study APN-002 of AD036 in OSA, as follows:

- In Study APN-002 efficacy of AD036 in reducing key measures of OSA severity including apnea-hypopnea index (AHI) and oxygen desaturation index (ODI) was correlated with certain patient baseline characteristics including those assessed by polysomnography (PSG). Study APN-006 will confirm this finding by enrolling patients from Study APN-002 who have baseline characteristics that predict increased responsiveness to AD036. New patients not previously screened in Study APN-002 who meet these criteria can also be enrolled in Study APN-006.
- There was evidence that the higher-dose formulation of AD036 (atomoxetine 75 mg/oxybutynin 5 mg) in Study APN-002 was superior to formulations of AD036 composed of lower dose combinations of atomoxetine and oxybutynin. However, comparison was not made of the combination of atomoxetine and oxybutynin to the individual components (i.e. atomoxetine alone or oxybutynin alone) which would more clearly establish the contribution of each component drug to the efficacy of the combination. Study APN-006 will compare the efficacy of AD036 (composed of commercially available formulations of atomoxetine 80 mg and oxybutynin 5 mg) in OSA to the efficacy of atomoxetine 80 mg alone and to placebo, in a three-period single-dose crossover design.

# 2.2 Background

# 2.2.1 Obstructive Sleep Apnea

The National Commission on Sleep Disorders Research identified sleep disorders as a major public health burden. OSA is the most common and serious of these sleep disorders and affects approximately 20 million people in the United States (US), with approximately 13% of men and 6% of women affected (Peppard et al, 2013). OSA is characterized by repetitive collapse or 'obstruction' of the pharyngeal airway during sleep, manifesting as repetitive episodes of hypopnea (i.e., shallow breathing) or apnea (i.e., paused breathing). These episodes of hypopnea or apnea may lead to arousal from sleep, sleep fragmentation, excessive daytime sleepiness, and/or neuropsychological impairment.

Research has shown that a number of pathogenic factors, or traits, contribute to the development of OSA (Eckert et al, 2013; Wellman et al, 2011; Wellman et al, 2013; Younes, 2003). The most important factors are the presence of an anatomically small, collapsible upper airway and a loss of pharyngeal muscle tone or responsiveness during sleep.

Long-term, OSA is associated with increased mortality and a number of adverse cardiovascular, neurocognitive, metabolic, and daytime functional consequences (Somers et al, 1995; Nieto et al, 2000; Brooks et al, 1997; Peppard et al, 2000; Hung et al, 1990; Wessendorf et al, 2000; Hoffstein, 1994; Shahar et al, 2001; Redline et al, 1997; Findley et al, 1988).

#### 2.2.2 Unmet Medical Need

Treatment for OSA has changed little over the past 40 years, with the overwhelming majority of patients treated with positive airway pressure, the most common of which is continuous positive airway pressure (CPAP), provided by a machine that mechanically maintains an open airway. Other treatments, such as pharyngeal surgery, mandibular advancement devices, and implantable nerve stimulators, were developed to address the anatomical predisposition to collapse; however, they have shown limited efficacy for niche populations.

While CPAP and related therapies are effective in improving sleep characteristics and oxygenation, many, perhaps most, patients find these devices uncomfortable or intolerable, and most estimates indicate that fewer than 50% of patients prescribed CPAP use it more than 4 hours per night, if at all (Weaver and Sawyer, 2010). Efforts to develop pharmacologic therapies, such as antidepressants, stimulants, and hormonal agents, for the treatment of OSA have been ongoing for at least 20 years, with no success thus far.

As many patients cannot use CPAP because they find it intolerable, this represents a significant health concern, as OSA is associated with numerous co-morbidities and increased mortality. Alternative options, such as drugs that activate the pharyngeal muscles are needed.

# 2.2.3 Biological Rationale

AD036 is a new fixed dose drug combination of atomoxetine and oxybutynin being developed for OSA. Atomoxetine is a pre-synaptic norepinephrine reuptake inhibitor indicated for the treatment of attention deficit hyperactivity disorder in children and adults. Oxybutynin is an antispasmodic drug that inhibits the muscarinic action of acetylcholine on smooth muscle and is indicated for the treatment of symptoms of bladder instability associated with voiding in patients with uninhibited neurogenic or reflex neurogenic bladder such as urgency, frequency, urinary leakage, urge incontinence and dysuria.

Efficacy and safety of AD036 for the signs and symptoms of OSA was recently evaluated in Apnimed's Phase 2 Study APN-002. There was evidence from this study that the high-dose

formulation of AD036 (atomoxetine 75 mg/oxybutynin 5 mg) was superior to formulations of AD036 composed of lower dose combinations of atomoxetine and oxybutynin, and to placebo. Efficacy of AD036 in OSA was correlated with certain patient baseline characteristics including those assessed by PSG. Study APN-006 will confirm and extend these findings by enrolling patients from Study APN-002 who have baseline characteristics that predict increased responsiveness to AD036. New patients not previously screened in Study APN-002 are also eligible for enrollment if all enrollment criteria are met.

# 3 Endpoints

| | Endpoints |
|---|---|
| Primary | Primary Efficacy Endpoint |
| | • AHI(4%), AD036 vs. placebo |
| Secondary | <ul> <li>Hypoxic burden and ODI(4%), AD036 vs. placebo</li> <li>Hypoxic burden, AHI(4%) and ODI(4%), AD036 vs. atomoxetine</li> </ul> |
| Tertiary | Tertiary Efficacy Endpoints |
| | • Total time with SaO2 <90% |
| | Snoring index |
| | • Sleep stages distribution and % of time in the various sleep stages |
| | Arousal index |
| | • Proportion of participants with ≥50% reduction, AHI and ODI endpoints |
| | • Fraction of hypopneas |
| | Alternative measures of AHI and ODI |
| Abbreviations: AHI = apr | nea-hypopnea index; ODI = oxygen desaturation index; SaO <sub>2</sub> = oxygen saturation. |

# 4 Study Design

# 4.1 Overall Design

Patients who participated in Study APN-002 are eligible for enrollment, as are new patients who meet enrollment criteria. A total of 54 patients who have baseline characteristics that, based on study 002 findings, predict increased responsiveness to AD036, will be planned for enrollment.

Objective OSA inclusion criteria for patients who participated in Study APN-002 will be determined based on the Study APN-002 baseline PSG exam (applies also to patients who were screened but did not meet the study PSG criteria). Objective OSA inclusion criteria for new patients can be based on a previous full night PSG or HSAT conducted at the site within 4 months prior to enrollment. If such results are not available, a screening HSAT may be conducted during the screening period, but such testing generally should be limited to patients with

documented previous sleep apnea test results (e.g. previous sleep study outside 4-month window) indicating the patient is still likely to meet objective OSA study enrollment criteria.

There are 3 randomized crossover HSAT nights. Each HSAT night is followed by a 1-week washout period. Dosing of the study treatment will occur immediately prior to bedtime. Patients will be randomized to treatment sequence with one of the following experimental treatments on each HSAT night:

- Atomoxetine 80 mg + oxybutynin 5 mg
- Atomoxetine 80 mg + placebo
- Placebo + placebo

Site personnel will contact participants remotely via telephone or video-call each HSAT night to assist with HSAT equipment use and to confirm study drug dosing.

Participants will be contacted by the site via telephone or video-call during each washout period to collect AE/SAE and concomitant medication information.

Overall study duration will be up to 10 weeks. Participants who withdraw from the study will not be replaced. No subsequent open-label extension is planned following the study.

Figure 1: Overview of Study Design



HSAT = home sleep apnea test.

# 4.2 Scientific Rationale for Study Design

The completed Phase 2 Apnimed Study APN-002 provided evidence of efficacy and safety for AD036 in OSA. This Phase 2 clinical study will further examine the efficacy and safety of AD036 in patients with baseline characteristics thought to predict increased responsiveness to the drug.

#### 4.3 Justification for Dose

The dose of AD036 in this study is the same or similar to the doses used in previous clinical studies that provided support for both the safety and efficacy of AD036 in OSA.

The study uses a dose of 80 mg atomoxetine (either alone or in combination with 5 mg oxybutynin). Previous single-dose crossover studies of the PK, safety, and efficacy of AD036 have demonstrated that this dosing is safe and well tolerated in the single-dose crossover setting.

A detailed description of the chemistry, pharmacology, efficacy, and safety of AD036 is provided in the Investigator's Brochure.

# 4.4 End of Study Definition

A participant is considered to have completed the study if he/she has completed all phases of the study including the final End of Study evaluation or the last scheduled procedure shown in the Schedule of Activities (SoA).

The end of the study is defined as the date of the last evaluation of the last participant in the study or last scheduled procedure shown in the SoA for the last participant in the study globally.

# 5 Study Population

The study population will consist both of participants from Study APN-002 and new patients who meet all enrollment criteria.

Participants must be able to provide written consent and meet all the inclusion criteria and none of the exclusion criteria.

#### 5.1 Inclusion Criteria

Individuals are eligible to be included in this study only if all of the following criteria apply:

#### Age and Sex

- 1. Male or Female, between 25 to 65 years of age, inclusive, at the Screening Visit.
  - Patients who participated in the APN-002 study can be enrolled if over the age of 65 years of age, up to 67 years of age.
  - Patients who did not participate in the APN-002 study must be between 25 to 65 years of age at the Screening Visit.

# **Objective Disease Measures**

- 2. AHI 10 to <20, or AHI  $\ge 20$  if any one of the following criteria are met:
  - Fraction of hypopneas ( $F_{hypopnea}$ ) is >90% or
  - Mean oxygen desaturation of obstructive events is  $\leq 4\%$  or
  - Fraction of hypopneas is 50-90% and mean oxygen desaturation is 4-8%

Note: Hypopneas defined by 4% oxygen desaturation

# Weight

3. BMI between 18.5 and 40 kg/m<sup>2</sup>, inclusive.

#### Male participants:

4. If male and sexually active with female partner(s) of childbearing potential, participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception (see Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information).

#### Female participants:

5. If a woman of childbearing potential (WOCBP), the participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception (See Appendix 4: Contraceptive Guidance and Collection of Pregnancy

- Information). All WOCBP must have negative result of a serum pregnancy test performed at screening.
- 6. If female and of non-childbearing potential, the participant must be either postmenopausal (defined as age ≥ 55 years with no menses for 12 or more months without an alternative medical cause) or permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

#### **Informed Consent**

- 7. Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the study-specific Screening Visit procedures.
- 8. Participant must be able to understand the nature of the study and must have the opportunity to have any questions answered.

#### 5.2 Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

# **Medical Conditions**

- 1. History of narcolepsy.
- 2. Clinically significant craniofacial malformation.
- 3. Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control. A medication for these purposes is defined by dosage form, such that a combination antihypertensive medication is considered 1 medication.
- 4. Clinically significant neurological disorder, including epilepsy/convulsions.
- 5. History of schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) or current International Classification of Disease criteria.
- 6. History of attempted suicide or suicidal ideation within 1 year prior to screening, or current suicidal ideation.
- 7. History of clinically significant constipation, gastric retention, or urinary retention.
- 8. Medically unexplained positive screen for drugs of abuse (excluding THC/marijuana) or substance use disorder as defined in DSM-V within 24 months prior to Screening Visit.
- 9. A significant new illness or infection requiring medical treatment in the past 30 days.

15 September 2020 13 of 45 V3.0

- 10. Clinically significant cognitive dysfunction.
- 11. Untreated narrow angle glaucoma.
- 12. Women who are pregnant or nursing.

#### **Prior/Concomitant Therapy**

- 13. CPAP should not be used for at least 2 weeks prior to first study HSAT.
- 14. History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.
- 15. History of using devices to affect participant sleeping position for the treatment of OSA, e.g. to discourage supine sleeping position, may enroll as long as the devices are not used during participation in the study.
- 16. History of oxygen therapy.
- 17. Use of medications from the list of disallowed concomitant medications during study participation.
- 18. Treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors, strong cytochrome P450 2D6 (CYP2D6) inhibitors, or monoamine oxidase inhibitors (MAOI) within 14 days of the start of treatment, or concomitant with treatment.

#### **Prior/Concurrent Clinical Study Experience**

19. Use of another investigational agent within 30 days or 5 half-lives prior to dosing, whichever is longer.

#### **Diagnostic Assessments**

20. Hepatic transaminases >2X the upper limit of normal (ULN), total bilirubin >1.5X ULN (unless confirmed Gilbert syndrome), estimated glomerular filtration rate < 60 ml/min.

#### **Other Exclusions**

- 21. <5 hours typical sleep duration.
- 22. Smoking more than 10 cigarettes or 2 cigars per day.
- 23. Unwilling to use specified contraception.
- 24. Unwilling to limit alcohol consumption to no greater than 2 units/day or less for men, or 1 unit/day for women, not to be consumed within 3 hours of bedtime.
- 25. Unwilling to limit caffeinated beverage intake (e.g., coffee, cola, tea) to 400 mg/day or less of caffeine, not to be used within 3 hours of bedtime.

15 September 2020 14 of 45 V3.0

- 26. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.
- 27. Participant considered by the investigator, for any reason, an unsuitable candidate to receive AD036 or unable or unlikely to understand or comply with the dosing schedule or study evaluations, including ability to use HSAT device.

# 5.3 Meals and Dietary Restrictions

- 1. Participants should refrain from consumption of any nutrients known to modulate CYP enzyme activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, pomegranate, and Seville or Moro [blood] orange products) within 72 hours before the first administration of study drug, during the study, and until final discharge.
- 2. Diet should be generally stable during the study, e.g., new diet programs should not be initiated.

# 5.4 Activity

There are no restrictions on physical activity during the study other than that physical activity should be generally stable during the study (e.g., new exercise programs should not be initiated).

#### 5.5 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently randomized to study treatment/entered into the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants that meets the Consolidated Standards of Reporting Trials publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any serious adverse events (SAEs).

Individuals who do not meet the criteria for participation in this study (screen failure) will not be rescreened, except if the opportunity for rescreening has been enabled by protocol amendment.

# **6 Study Treatment**

Study treatment is defined as any investigational treatment(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

# **6.1 Study Treatments**

Study treatments include atomoxetine, oxybutynin, and placebo, taken immediately before the participant's planned bedtime on HSAT nights, in randomized order:

15 September 2020 15 of 45 V3.0

- Atomoxetine 80 mg + oxybutynin 5 mg
- Atomoxetine 80 mg + placebo
- Placebo + placebo

| Study Treatment Name: | Atomoxetine<br>hydrochloride | Oxybutynin chloride | Placebo<br>(Microcrystalline<br>Cellulose) |
|---|---|---|---|
| <b>Dosage Formulation:</b> | Capsule | Tablet | Capsule |
| Dosage Level: | 80 mg | 5 mg | 250mg |
| Route of Administration: | Oral | Oral | Oral |
| <b>Dosing Instructions:</b> | 1 capsule<br>administered with<br>water | 1 tablet<br>administered with<br>water | 1 tablet<br>administered with<br>water |
| Storage/Packaging/Labeling: | Store per package insert. | Store per package insert. | Controlled room temperature. |

# 6.2 Preparation/Handling/Storage/Accountability

- Only participants enrolled in the study may receive study treatments. Prior to
  distribution to participants all study treatments must be stored in a secure,
  environmentally controlled, and monitored (manual or automated) area in accordance
  with the labeled storage conditions with access limited to the Investigator and
  authorized site staff.
- The Investigator, institution, or the head of the medical institution (where applicable) is responsible for study treatment accountability, reconciliation, and record maintenance (i.e., receipt, reconciliation, and final disposition records).
- After receiving Sponsor approval in writing, sites are responsible for returning all
  unused or partially used study treatment to the Sponsor or designated third party or for
  preparing the study treatment for destruction via incineration.
- Returned study treatment should not be re-dispensed to participants

#### **6.3** Measures to Minimize Bias

All participants will be centrally randomized for the crossover study. Each participant will be assigned a unique number (randomization number) that encodes the participant's assignment to one of the sequences of the study, according to the randomization schedule using a validated computer program.

# **6.4 Study Treatment Compliance**

Participants will be required to return any unused study drug. Unused study drug will be counted and recorded by study personnel to assess study treatment compliance.

# 6.5 Concomitant Therapy

Concomitant therapy with the following medications is disallowed:

- MAOIs or other drugs that affect monoamine concentrations (e.g., rasagiline) [MAOIs are contraindicated for use with atomoxetine]
- Selective Serotonin Reuptake Inhibitors (e.g., paroxetine)
- Selective Norepinephrine Reuptake Inhibitors (e.g., duloxetine)
- Norepinephrine Reuptake Inhibitors (e.g., reboxetine)
- Alpha-1 antagonists (e.g., tamsulosin)
- Tricyclic antidepressants (e.g., desipramine)
- Centrally acting antihypertensives (e.g. clonidine, alpha-methyl-DOPA)
- CYP2D6 inhibitors
- Strong CYP3A4 inhibitors (e.g., ketoconazole)
- Benzodiazepines and other anxiolytics
- Opioids
- Sedative hypnotics
- Muscle relaxants
- Pressor agents
- Drugs with clinically significant cardiac QT-interval prolonging effects
- Drugs known to lower seizure threshold (e.g., chloroquine)
- Amphetamines
- Antiepileptics
- Antiemetics
- Modafinil or armodafinil
- Beta<sub>2</sub> agonists (e.g., albuterol)

- Antipsychotics
- Anticholinergics and anticholinesterase inhibitors, including drugs with substantial anticholinergic side effects, (e.g., first generation antihistamines)
- Sedating antihistamines
- Pseudoephedrine, phenylephrine, oxymetazoline
- Nicotine replacement products
- Most drugs for Parkinson's, Alzheimer's, Huntington's, Amyotrophic Lateral Sclerosis, or drugs for other neurodegenerative diseases

Medications that do not have substantial effects on the central nervous system (CNS), respiration, or muscle activity are generally allowed if dose and frequency is stable<sup>2</sup> for 1 month prior to enrollment and during the course of the study, including, but not necessarily limited to, the following drugs and drug classes:

- Non-centrally acting antihypertensives (angiotensin-converting-enzyme/angiotensin II receptor blocker inhibitors, calcium channel blockers, spironolactone, hydrochlorothiazide, etc.)
- Statins
- Proton pump inhibitors and histamine h<sub>2</sub> receptor blockers
- Over-the-counter (OTC) antacids
- Non-sedating antihistamines (e.g., cetirizine, loratadine)
- Melatonin
- Non-steroidal anti-inflammatory drugs and acetaminophen
- Laxatives
- Erectile dysfunction drugs
- Inhaled corticosteroids (e.g., fluticasone)
- Antidiabetics
- Ocular hypotensives and other ophthalmics (e.g., timolol)
- Hormonal therapy (e.g., estrogen replacement or anti-estrogens) and hormonal contraceptives

15 September 2020 18 of 45 V3.0

<sup>&</sup>lt;sup>2</sup> Drugs that are used intermittently are considered to be used at a stable dose and frequency if the general pattern of use over time is consistent with the patient's previous use.

- Thyroid medications
- Anticoagulants
- OTC topicals (e.g., topical pain relievers)
- Osteoporosis drugs

# 6.6 Treatment After the End of the Study

Not applicable. No subsequent open-label extension is planned following the study. Study treatment will not be available after the end of study participation.

# 7 Discontinuation of Study Treatment

If a clinically significant finding is identified, the Investigator or qualified designee will determine if the participant can continue in the study and if any change in participant management is needed. Any new clinically relevant finding should be reported as an adverse event (AE).

# 7.1 Stopping Criteria

# 7.1.1 Individual Participant Stopping Criteria

- Incidents of abuse, diversion, or misuse of the study treatment.
- Incidents of clinical significance: hallucinations, amnesia, delusional thinking, delirium, manic symptoms, aggressive behavior, suicidality, homicidality, agitation, confusion, or convulsions/seizures.
- Participants reporting any SAE.
- Acute urinary obstruction.
- Any other AE that in the judgment of the Investigator necessitates the participant stopping to protect participant safety.

# 7.2 Participant Discontinuation/Withdrawal from the Study

- A participant may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the Investigator for safety, behavioral, or administrative reasons.
- If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.

- If a participant withdraws from the study, he/she may request destruction of any samples taken and not tested, and the Investigator must document this in the site study records.
- All participants who withdraw from the study with an ongoing AE must be followed until the event is resolved or deemed stable.
- Participation may be terminated before completing the study and the reason recorded.

# 7.3 Loss of Participants to Follow-Up

A participant will be considered lost to follow-up if the study site is repeatedly unable to contact the participant. The following actions must be taken if a participant is lost to follow-up:

- The site must attempt to contact the participant and resume study activities as soon as possible (and within the activity window, where one is defined) and counsel the participant on the importance of maintaining the assigned activity schedule and ascertain whether or not the participant wishes to and/or should continue in the study.
- In cases in which the participant is deemed lost to follow-up, the Investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record/eCRF.
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

# 8 Study Assessments and Procedures

- Study procedures and their timing are summarized in the SoA.
- Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential
  participants meet all eligibility criteria. The Investigator will maintain a screening log to
  record details of all participants screened and to confirm eligibility or record reasons for
  screening failure, as applicable.

15 September 2020 20 of 45 V3.0

# 8.1.1 Home Sleep Apnea Testing (HSAT)

- Methods: Standard HSAT recording and data interpretation will be performed in accordance
  with the American Academy of Sleep Medicine (AASM) scoring manual for respiratory
  signals. EEG activity will be estimated from frontal derivations. Screening HSAT for new
  patients may be conducted without estimation of EEG activity.
- Time of lights out will be according to the participants' habitual schedule and kept constant across the HSAT study nights.
- Sites will instruct participants on proper use of HSAT device at screening visit.
- Sites will contact participants each night of study drug dosing to assist and confirm use of HSAT and study drug dosing.
- Scoring: For uses other than establishing that the patients meets study enrollment criteria, all HSATs will be scored by centralized technologists who are separate from the clinical care team.

# 8.2 Safety Assessments

- Planned time points for all adverse events assessments are provided in the SoA.
- Safety monitoring will be guided by the established safety profiles of atomoxetine and oxybutynin, and by Phase 1 and 2 safety data for the combination, and will include monitoring and recording of AEs, SAEs, and recording of study or treatment discontinuations. Effects on OSA will also be monitored by HSAT.

#### **8.3** Adverse Events and Serious Adverse Events

The definitions of AEs and SAEs can be found in Appendix 3.

Adverse events will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).

The Investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up on AEs that are serious, considered related to the study treatment or the study, or that caused the participant to discontinue the study and/or study treatment (see Section 7).

# 8.3.1 Time Period and Frequency for Collecting AE and SAE Information

All AEs and SAEs will be collected from the signing of informed consent form (ICF) until the end of the study.

All SAEs will be recorded and reported to the Sponsor or designee within 24 hours. The Investigator will submit any updated SAE data to the Sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek AEs or SAEs after the conclusion of study participation. However, if the Investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study treatment or study participation, the Investigator must promptly notify the Sponsor.

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3.

# 8.3.2 Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about AE occurrence.

# 8.3.3 Follow-up of AEs and SAEs

After the initial AE/SAE report, the Investigator is required to proactively follow each participant at subsequent contacts. All SAEs will be followed until resolution, stabilization, until the event is otherwise explained, or the participant is lost to follow-up. Further information on follow-up procedures is given in Appendix 3.

# **8.3.4** Regulatory Reporting Requirements for SAEs

- Prompt notification (within 24 hours, see Appendix 3) by the Investigator to the Sponsor of an SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study treatment under clinical investigation are met.
- The Sponsor has a legal responsibility to notify both the local regulatory authority and other
  regulatory agencies about the safety of a study treatment under clinical investigation. The
  Sponsor will comply with country-specific regulatory requirements relating to safety
  reporting to the regulatory authority, IRB/Independent Ethics Committees (IEC), and
  Investigators.
- Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and Sponsor policy and forwarded to Investigators as necessary.

15 September 2020 22 of 45 V3.0

 An Investigator who receives an Investigator safety report describing an SAE or other specific safety information (e.g., summary or listing of SAE) from the Sponsor will file it along with the Investigator's Brochure and will notify the IRB/IEC, if appropriate according to local requirements.

# 8.3.5 Pregnancy

- Details of all pregnancies in female participants after the start of study treatment and until at least 5 terminal half-lives after the last dose will be collected.
- If a pregnancy is reported, the Investigator should inform the Sponsor within 24 hours of learning of the pregnancy and should follow the procedures outlined in Appendix 4.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered to be SAEs.

# **8.4** Treatment of Overdose

For this study, any dose of atomoxetine greater than 80 mg and of oxybutynin greater than 5 mg more frequently than QHS will be considered an overdose.

In the event of an overdose, the Investigator should refer to the approved product labels for atomoxetine and oxybutynin for advice on overdose and:

- 1. Document the quantity of the excess dose as well as the duration of the overdosing in the eCRF.
- 2. Contact the Medical Monitor.
- 3. Closely monitor the participant as clinically indicated for AE/SAE and laboratory abnormalities until atomoxetine and/or oxybutynin can no longer be detected systemically.
- 4. Obtain a plasma sample for PK analysis, if clinically indicated, within 1 day from the date of the last dose of study treatment if requested by the Medical Monitor (determined on a case by case basis).

Decisions regarding dose interruptions or modifications will be made by the Investigator in consultation with the Medical Monitor based on the clinical evaluation of the participant.

#### 8.5 Pharmacokinetics

PK parameters are not evaluated in this study.

15 September 2020 23 of 45 V3.0

# 9 Statistical Considerations and Sample Size Determination

The efficacy of AD036 in OSA was investigated in Apnimed Study APN-002. Patients in Study APN-006 will be selected based on baseline objective OSA criteria that, from the results of Study APN-002, are thought to enrich for patients more likely to be responders. A total of 54 patients (9 per sequence) will enter the 3-treatment crossover study. The study will have 90% power to detect a treatment difference at a two-sided 0.05 significance level, if the true difference between treatments on AHI is -11.000 units. This assumes that the within-subject standard deviation is 12, estimated from Study APN-002 using a subset of 92 subjects with baseline  $F_{hypopnea} \ge 65\%$ .

Subjects will be randomized to one of the following 6 sequences: A - B - C, B - C - A, C - B - A, A - C - B, B - A - C, C - A - B. This design is both uniform within sequences (each treatment appears the same number of times within each sequence) and uniform within periods (each treatment appears the same number of times within each period). These properties result in neither the sequence nor the period effects being aliased with the treatment effect. Furthermore, the inclusion of a washout period is believed to minimize any carryover effect, or at the minimum, the carryover effect is believed to be equal among all treatments and therefore would not be aliased with the estimation of the treatment effect. The above design also assures that each treatment is preceded by all other treatments at least once.

# 9.1 Populations for Analyses

For the purposes of analysis, the following analysis sets are defined:

| Population | Description |
|---|---|
| Enrolled | All participants who signed the ICF (including screening failures). |
| Modified Intent to Treat (mITT) Population | The mITT Population comprises all participants who take at least 1 dose of any of the study treatments, and have at least 1 measurement on the primary endpoint. Participants will be analyzed for efficacy according to the treatment group into which they are randomized. |
| Safety Population | The Safety Population consists of all participants who are randomized and receive at least 1 dose of any of the study treatments. Participants will be analyzed for safety based on the treatment received. A precise definition of "as actually received" will be added in the Statistical Analysis Plan (SAP). |
| Per Protocol (PP) Population | The PP Population consists of all participants without any major protocol violations that could influence efficacy assessment, and who are compliant with the study medication and HSAT in each crossover period. Participants in this population will be analyzed according to the treatment they actually received. |

# 10 Supporting Documentation and Operational Considerations

# 10.1 Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

# 10.1.1 Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organizations of Medical Sciences International Ethical Guidelines.
  - Applicable International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines.
  - o Applicable laws and regulations.
- The protocol, protocol amendments, ICF, Investigator's Brochure, and other relevant documents (e.g., advertisements) must be submitted to an IRB/IEC by the Investigator and reviewed and approved by the IRB/IEC before the study is initiated.
- The Investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC.
- Notifying the IRB/IEC of SAE or other significant safety findings as required by IRB/IEC procedures.
- Overall conduct of the study at the site and adherence to requirements of 21 Code of Federal Regulations (CFR), ICH GCP guidelines, the IRB/IEC guidelines, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations.

#### **10.1.2** Financial Disclosure

Investigators and sub-Investigators will provide the Sponsor with sufficient, accurate financial information in accordance with local regulations to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### **10.1.3 Informed Consent Process**

- The Investigator or his/her representative will explain the nature of the study to the participant or his/her legally authorized representative and answer all questions regarding the study.
- Participants must be informed that their participation is voluntary. Participants will be
  required to sign a statement of informed consent that meets the requirements of 21 CFR 50,
  local regulations, ICH guidelines, Health Insurance Portability and Accountability Act
  requirements, where applicable, and the IRB/IEC or study center.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Participants must be re-consented to the most current version of the ICF(s) during their participation in the study.
- A copy of the signed ICF(s) must be provided to the participant or the participant's legally authorized representative.

15 September 2020 26 of 45 V3.0

• If a protocol amendment is required, the ICF may need to be revised to reflect the changes to the protocol. If the ICF is revised, it must be reviewed and approved by the appropriate IEC/IRB, and signed by all participants subsequently enrolled in the study as well as those currently enrolled in the study.

#### 10.1.4 Data Protection

- Participants will be assigned a unique identifier by the Sponsor. Any participant records or datasets that are transferred to the Sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the Sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant.
- The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the Sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

# 10.1.5 Dissemination of Clinical Study Data

When the clinical study report is completed, the Sponsor will provide the major findings of the study to the Investigator. A summary of the study results will also be posted in a publicly accessible database (e.g., www.ClinTrials.gov). The results may also be submitted for publication.

# **10.1.6 Data Quality Assurance**

- All participant data relating to the study will be recorded on printed or eCRFs unless transmitted to the Sponsor or designee electronically. The Investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF.
- The Investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.
- The Investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory agency inspections and provide direct access to source data documents.
- The Sponsor or designee is responsible for the data management of this study including quality checking of the data.

15 September 2020 27 of 45 V3.0

- Study monitors will perform ongoing source data verification to confirm that data entered into the eCRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.
- Records and documents, including signed ICF, pertaining to the conduct of this study must be
  retained by the Investigator for 5 years after study completion unless local regulations or
  institutional policies require a longer retention period. No records may be destroyed during
  the retention period without the written approval of the Sponsor. No records may be
  transferred to another location or party without written notification to the Sponsor.
- All data generated by the site personnel will be captured electronically at each study center using eCRFs. Once the eCRF clinical data have been submitted to the central server at the independent data center, corrections to the data fields will be captured in an audit trail. The reason for change, the name of the person who performed the change, together with the time and date will be logged to provide an audit trail.
- If additional corrections are needed, the responsible monitor or data manager will raise a query in the electronic data capture (EDC) application. The appropriate staff at the study site will answer queries sent to the Investigator. The name of the staff member responding to the query, and time and date stamp will be captured to provide an audit trail. Once all source data verification is complete and all queries are closed, the monitor will lock the database.
- The specific procedures to be used for data entry and query resolution using the EDC system/eCRF will be provided to study sites in a training manual. In addition, site personnel will receive training on the EDC system/eCRF.

#### **10.1.7** Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the Investigator's site.
- Data entered in the eCRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The Investigator may need to request previous medical records or transfer records, depending on the study.
- Definition of what constitutes source data can be found in Section 10.1.11.1.

15 September 2020 28 of 45 V3.0

# 10.1.8 Study and Site Closure

The Sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the Sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study site closure evaluation has been performed.

The Investigator may initiate study site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the Sponsor or Investigator may include but are not limited to:

- Failure of the Investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the Sponsor's procedures, or GCP guidelines.
- Inadequate recruitment of participants by the Investigator.
- Discontinuation of further study treatment development.

# **10.1.9 Publication Policy**

- The sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data.
- Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.
- The Sponsor retains the right to disapprove any submission for publication, including any publication using trial data, including abstracts, presentations or manuscripts.

# 10.1.10 Protocol Approval and Amendment

Before the start of the study, the study protocol and/or other relevant documents will be approved by the IEC/IRB/Competent Authorities, in accordance with local legal requirements. The Sponsor must ensure that all ethical and legal requirements have been met before the first participant is enrolled in the study.

This protocol is to be followed exactly. To alter the protocol, amendments must be written, receive approval from the appropriate personnel, and receive IRB/IEC/Competent Authority approval prior to implementation (if appropriate). Following approval, the protocol amendment(s) will be submitted to the US Investigational New Drug (IND) under which the study is being conducted.

Administrative changes (not affecting the participant benefit/risk ratio) may be made without the need for a formal amendment. All amendments will be distributed to all protocol recipients, with appropriate instructions.

# 10.1.11 Liability and Insurance

The Sponsor will take out reasonable third-party liability insurance cover in accordance with all local legal requirements. The civil liability of the Investigator, the persons instructed by him or her and the hospital, practice, or institute in which they are employed and the liability of the Sponsor with respect to financial loss due to personal injury and other damage that may arise as a result of the carrying out of this study are governed by the applicable law.

The Sponsor will arrange for participants participating in this study to be insured against financial loss due to personal injury caused by the pharmaceutical products being tested or by medical steps taken in the course of the study.

# 10.1.11.1 Access to Source Data

During the study, a monitor will either make site visits or request documentation remotely to review protocol compliance, compare EDC/eCRF entries and individual participant's medical records, assess drug accountability, and ensure that the study is being conducted according to pertinent regulatory requirements. The EDC/eCRF entries will be verified with source documentation. The review of medical records will be performed in a manner to ensure that participant confidentiality is maintained.

Checking of the EDC/eCRF entries for completeness and clarity, and cross-checking with source documents, will be required to monitor the progress of the study. Moreover, regulatory authorities of certain countries, IRBs, IECs, and/or the Sponsor's Clinical Quality Assurance Group may wish to carry out such source data checks and/or on-site audit inspections. Direct access to source data will be required for these inspections and audits; they will be carried out giving due consideration to data protection and medical confidentiality. The Investigator assures the CRO and the Sponsor of the necessary support at all times.

# **10.2 Appendix 2: Clinical Laboratory Tests**

- Protocol-specific requirements for inclusion or exclusion of participants are detailed in Section 5 of the protocol.
- Laboratory testing is performed non-fasting.
- Additional tests may be performed at any time during the study as determined necessary by the Investigator or required by local regulations.

15 September 2020 30 of 45 V3.0

**Table 2: Protocol-Required Safety Laboratory Assessments** 

| Laboratory<br>Assessments | Parameters | | |
|---|---|---|---|
| Hematology | Hematocrit Hemoglobin Platelet Count RBC Count | RBC Indices | WBC count with Differential |
| Serum Chemistry | Albumin BUN Creatinine Potassium Sodium Bilirubin Total Protein | ALT AST Alkaline phosphatase Calcium Glucose Chloride Bicarbonate | |
| Routine<br>Urinalysis | Specific gravity pH, protein (albumin), glucose, ketones, blood (RBC), WBC by dipstick Microscopic examination (if blood or protein is abnormal) | | |
| Other Tests | <ul> <li>CYP 2D6 (only at Screening Visit, only for new patients not previously tested in Study 002)</li> <li>HbA1c (Screening Visit only)</li> <li>Serum hCG pregnancy test at screening. Additional testing may be performed if needed in WOCBP.</li> <li>Urine drugs of abuse (marijuana, cocaine, amphetamine, methamphetamine, opiates, phencyclidine)</li> </ul> | | |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen; CYP2D6 = cytochrome P450 2D6; γ-GTP = gamma guanosine-5'-triphosphate; HbA1c = hemoglobin A1c (glycated hemoglobin); hCG = human chorionic gonadotropin; MCH = mean corpuscular hemoglobin; MCV = mean corpuscular volume; RBC = red blood cell count; WBC= white blood cell; WOCBP = women of childbearing potential.

Investigators must document their review of each laboratory safety report.

# 10.3 Appendix 3: AE Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### **Definition of AE**

#### **AE Definition**

- An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the medicinal product.
- NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or
  other safety assessments (e.g., ECG, radiological scans, vital signs measurements),
  including those that worsen from baseline, considered clinically significant in the medical
  and scientific judgment of the Investigator (i.e., not related to progression of underlying
  disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study treatment administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study treatment or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.
- "Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as an AE or SAE if they fulfill the definition of an AE or SAE.

# **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments which are associated with the underlying disease, unless judged by the Investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### **Definition of SAE**

If an event is not an AE per definition above, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

## An SAE is defined as any untoward medical occurrence that, at any dose:

#### Results in death

#### Is life-threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AE. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

# Results in persistent disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### Is a congenital anomaly/birth defect

#### Other situations

• Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical treatment to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.

Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

#### Recording and Follow-up of AE and SAE

#### **AE and SAE Recording**

- When an AE/SAE occurs, it is the responsibility of the Investigator to review all documentation (e.g., hospital progress notes, laboratory, and diagnostics reports) related to the event.
- The Investigator will then record all relevant AE/SAE information in the eCRF.
- It is **not** acceptable for the Investigator to send photocopies of the participant's medical records in lieu of completion of the AE/SAE eCRF page.
- There may be instances when copies of medical records for certain cases are requested by the CRO's. In this case, all participant identifiers, with the exception of the participant number, will be blinded on the copies of the medical records before submission to the CRO's Clinical Studies Safety Center.

15 September 2020 34 of 45 V3.0

• The Investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. In such cases, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### **Assessment of Intensity**

The Investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to one of the following categories:

- Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event; and both AE and SAE can be assessed as severe.

An event is defined as 'serious' when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

# **Assessment of Causality**

- The Investigator is obligated to assess the relationship between study treatment and each occurrence of each AE/SAE.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The Investigator will use clinical judgment to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study treatment administration will be considered and investigated.
- The Investigator will also consult the Investigator's Brochure and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the Investigator <u>must</u> document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.

15 September 2020 35 of 45 V3.0

- There may be situations in which an SAE has occurred and the Investigator has minimal information to include in the initial report to the CRO. However, it is very important that the Investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the CRO.
- The Investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-up of AE and SAE

- The Investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the CRO to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- If a participant dies during participation in the study the Investigator will provide the CRO with a copy of any post-mortem findings including histopathology.
- New or updated information will be recorded in the originally completed eCRF.
- The Investigator will submit any updated SAE data to the CRO within 24 hours of receipt of the information.

#### **Reporting of SAE to CRO**

# SAE Reporting to CRO Via EDC Tool

- The Investigator must report any SAEs to the CRO within 24 hours of becoming aware of the event.
- When calling to report an SAE, state that you are reporting an SAE and give the Investigator's name, your name, the telephone number where you can be reached, and the protocol number and title.

15 September 2020 36 of 45 V3.0

- The Investigator and the Sponsor (or Sponsor's designated agent) will review each SAE report and the Sponsor/CRO will evaluate the seriousness and the causal relationship of the event to study treatment. In addition, the Sponsor (or Sponsor's designated agent) will evaluate the expectedness according to the reference documents (Investigator's Brochure or US product labeling for atomoxetine or oxybutynin). Based on the Investigator and Sponsor's assessment of the event, a decision will be made concerning the need for further action.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form (see next section) or by telephone.
- Contacts for SAE reporting can be found in the Study Reference Manual.

All SAEs will be recorded from signing of informed consent until the end of the study as defined in Section 4.4. Serious adverse events occurring after the end of the study and coming to the attention of the Investigator must be reported only if they are considered (in the opinion of the Investigator) causally-related to study treatment.

#### **Suspected Unexpected Serious Adverse Reactions (SUSARs)**

Any AE that is serious, associated with the use of the study treatment, and unexpected (SUSAR) has additional reporting requirements, as described below.

- If the SUSAR is fatal or life-threatening, associated with study treatment, and unexpected, regulatory authorities and IECs will be notified within 7 calendar days after the Sponsor learns of the event. Additional follow-up (cause of death, autopsy report, and hospital report) information should be reported within an additional 8 days (15 days total).
- If the SUSAR is not fatal or life-threatening but is otherwise serious, associated with study treatment, and unexpected, regulatory authorities and IECs will be notified within 15 calendar days after the Sponsor learns of the event.

The Sponsor will notify the Investigators in a timely fashion of relevant information about SUSARs that could adversely affect the safety of participants. Follow-up information may be submitted if necessary.

15 September 2020 37 of 45 V3.0

The Sponsor will also provide annual safety updates to the regulatory authorities and IECs responsible for the study. These updates will include information on SUSARs and other relevant safety findings.

# 10.4 Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information

#### **Definitions**

#### WOCBP

A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile (see below).

Women in the following categories are not considered WOCBP:

- 1. Premenarchal
- 2. Premenopausal female with one of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

NOTE: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

- 3. Post-menopausal female
  - A post-menopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the post-menopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
  - Females on HRT and whose menopausal status is in doubt will be required to use one of the non-estrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status before study enrollment.

# **Contraception Guidance:**

### **Male Participants:**

Male participants with female partners of childbearing potential are eligible to participate if they agree to ONE of the following during the protocol-defined time frame in Section 5.1:

- Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.
- Agree to use a contraceptive method with a failure rate of <1% per year as described in the table below when having penile-vaginal intercourse with a WOCBP who is not currently pregnant.

In addition, male participants must refrain from donating sperm for the duration of the study and for 3 months after the last dose of study treatment.

Male participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or to use a male condom during each episode of penile penetration during the protocol-defined time frame.

# **Female Participants**

Female participants of childbearing potential are eligible to participate if they agree to use a highly effective method of contraception consistently and correctly as described in the table below.

# Highly Effective Contraceptive Methods That Are User Dependent<sup>1</sup>

Failure rate of <1% per year when used consistently and correctly.

Combined (estrogen- and progestin-containing) hormonal contraception associated with inhibition of ovulation<sup>2</sup>

- Oral
- Intravaginal
- Transdermal

Progestogen-only hormonal contraception associated with inhibition of ovulation

- Oral
- Injectable

## Highly Effective Contraceptive Methods That Are User Independent<sup>1</sup>

Implantable progestogen-only hormonal contraception associated with inhibition of ovulation

- IUD
- Intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion

#### Vasectomized partner

A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### Sexual abstinence

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

#### NOTES:

1 Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies.

#### **Pregnancy Testing**

- WOCBP should only be included after a confirmed menstrual period. and a negative highly sensitive serum pregnancy test.
- Pregnancy testing will be performed whenever a menstrual cycle is missed or when pregnancy is otherwise suspected.

## Female participants who become pregnant

- The Investigator will collect pregnancy information on any female participant who becomes pregnant while participating in this study. Information will be recorded on the appropriate form and submitted to the Sponsor within 24 hours of learning of a participant's pregnancy. The participant will be followed to determine the outcome of the pregnancy. The Investigator will collect any follow up information on the participant and the neonate and the information will be forwarded to the Sponsor. Generally, follow up will not be required for longer than 6 to 8 weeks beyond the estimated delivery date. Any termination of the pregnancy will be reported, regardless of fetal state (presence or absence of anomalies) or indication for the procedure.
- While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or elective termination of a pregnancy will be reported as an AE or SAE. A spontaneous abortion is always considered to be an SAE and will be reported as such. Any post-study pregnancy-related SAE considered reasonably related to the study treatment by the Investigator will be reported to the Sponsor as described in Section 8.3.4. While the Investigator is not obligated to actively seek this information in former study participants, he or she may learn of an SAE through spontaneous reporting.
- Any female participant who becomes pregnant while participating in the study will be withdrawn from the study.

# 10.5 Appendix 5: List of Abbreviations

AHI apnea-hypopnea index

AE adverse event

BMI body mass index

CFR Code of Federal Regulations

CNS central nervous system

CPAP continuous positive air pressure

CSSA Cocaine Selective Severity Assessment

CYP2D6 cytochrome P450 2D6 CYP3A4 cytochrome P450 3A4

DSM-5 Diagnostic and Statistical Manual of Mental Disorders, 5th edition

ECG electrocardiogram

EEG electroencephalogram

eCRF electronic case report form(s)

EDC electronic data capture
ESS Epworth Sleepiness Scale
FSH follicle-stimulating hormone

GCP Good Clinical Practice

HRT hormone replacement therapy

HSAT Home sleep apnea test ICF informed consent form

ICH International Conference on Harmonisation

IEC Independent Ethics Committee

IND Investigational New Drug
IRB Institutional Review Board

IRT Interactive Response Technology

OSA obstructive sleep apnea

OTC over-the-counter

MAOI monoamine oxidase inhibitor NREM non-rapid eye movement

PGI-S Participant Global Impression of Severity

PK pharmacokinetic(s)
PSG polysomnography

DWRT Delayed Word Recall Test
QHS 1 dose every night at bedtime

| REM | rapid eye movement |
|-----|---------------------------|
| SAE | serious adverse event |
| SAP | Statistical Analysis Plan |
| SoA | Schedule of Activities |

SUSAR suspected unexpected serious adverse reaction

ULN upper limit of normal

US United States

WOCBP woman of childbearing potential

# 11 References

Brooks D, Horner RL, Kozar LF, Render-Teixeira CL, Phillipson EA. Obstructive sleep apnea as a cause of systemic hypertension. Evidence from a canine model. J Clin Invest 1997;99:106-109.

Chan E, Steenland HW, Liu H, Horner RL. Endogenous excitatory drive modulating respiratory muscle activity across sleep-wake states. Am J Respir Crit Care Med 2006;174:1264-1273.

Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med 2013;188:996-1004.

Findley LJ, Unverzagt ME, Suratt PM. Automobile accidents involving patients with obstructive sleep apnea. Am Rev Respir Dis 1988;138:337-340.

Hoffstein V. Blood pressure, snoring, obesity, and nocturnal hypoxaemia. Lancet 1994;344:643-645.

Hung J, Whitford EG, Parsons RW, Hillman DR. Association of sleep apnoea with myocardial infarction in men. Lancet 1990;336:261-264.

Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, et al. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA 2000; 283:1829-1836.

Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol 2013;177(9):1006–1014.

Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med 2000; 342:1378-1384.

Redline S, Strauss ME, Adams N, Winters M, Roebuck T, Spry K, et al. Neuropsychological function in mild sleep-disordered breathing. Sleep 1997; 20:160-167.

Shahar E, Whitney CW, Redline S, Lee ET, Newman AB, Nieto FJ, et al. Sleep-disordered breathing and cardiovascular disease: Cross-sectional results of the Sleep Heart Health Study. Am J Respir Crit Care Med 2001;163:19-25.

Somers VK, Dyken ME, Clary MP, Abboud FM. Sympathetic neural mechanisms in obstructive sleep apnea. J Clin Invest 1995;96:1897-1904.

Weaver TE, Sawyer AM. Adherence to continuous positive airway pressure treatment for obstructive sleep apnea: implications for future interventions. Indian J Med Res 2010;131:245-258.

Wellman A, Eckert DJ, Jordan AS, Edwards BA, Passaglia CL, Jackson AC, et al. A method for measuring and modeling the physiological traits causing obstructive sleep apnea. J Appl Physiol (1985) 2011; 110:1627-1637.

Wellman A, Edwards BA, Sands SA, Owens RL, Nemati S, Butler J, et al. A simplified method for determining phenotypic traits in patients with obstructive sleep apnea. J Appl Physiol (1985) 2013;114:911-922.

Wessendorf TE, Teschler H, Wang YM, Konietzko N, Thilmann AF. Sleep-disordered breathing among patients with first-ever stroke. J Neurol 2000;247:41-47.

Younes M. Contributions of upper airway mechanics and control mechanisms to severity of obstructive apnea. Am J Respir Crit Care Med 2003;168:645-658.

15 September 2020 44 of 45 V3.0

## **Declaration of the Investigator**

**Title:** Phase 2, Randomized, 3-Period, Placebo-Controlled Crossover Study to Evaluate the Efficacy and Safety in Obstructive Sleep Apnea of AD036 versus Placebo or Atomoxetine

All documentation for this study that is supplied to me and that has not been previously published will be kept in the strictest confidence. This documentation includes this study protocol, Investigator's Brochure, EDC system/eCRF, and other scientific data.

The study will not be commenced without the prior written approval of a properly constituted IRB or IEC. No changes will be made to the study protocol without the prior written approval of the Sponsor and the IRB or IEC, except where necessary to eliminate an immediate hazard to the participants.

I have read and understood and agree to abide by all the conditions and instructions contained in this protocol.

# Signature Name (block letters) Title (block letters) Institution (block letters) Phone number

Responsible Investigator of the local study center